CLINICAL TRIAL: NCT01817920
Title: Integrated Interdisciplinary Program for Fall Prevention in Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CCH-091237
Record Dates: First submitted 2013-03-20; First posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: the Fall Rates; the Severity of Injuries

ARMS (1):
- integrated multidisciplinary fall prevention program (Experimental)
  Interventions: Behavioral: integrated multidisciplinary fall prevention program

INTERVENTIONS:
Behavioral: integrated multidisciplinary fall prevention program

SUMMARY:
Falls are very common accidents in Hospital. It not only results in injuries, less mobility among patients but increases their length of stay, cost and family burdens. Reducing the rates and injuries of falls is an urgent issue around hospitals.

An integrated multidisciplinary fall prevention program (IMFPP) was implemented from 2006 in CCH. Members include physicians, nurses, case manager therapists, engineers and staffs of maintenance. The aim of this study is to determine whether IMFPP efforts support interventions with multiple components do reduce the fall rates and severity of injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patient in CCH's fall incidence reports system

Exclusion Criteria:

* No

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2004-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Severities of injury as fall | within 1 day after fall
  Severities of injury was according to Taiwan Quality Indicator Project (TQIP)
  1. mild injury (contusion, abrasion wound)
  2. moderate injury (sprain, laceration wound)
  3. severe injury (fracture, conscious loss)

SECONDARY OUTCOMES:
Rate of recurrent fall | participants will be followed for the duration of hospital stay, an expected average of 4 weeks